CLINICAL TRIAL: NCT04558151
Title: Randomized-controlled Trial of Spirometry-Assisted Preoperative INSPIRAtory Muscle Training on Postoperative Complications in Abdominal Surgery in a Single Tertiary Referral Centre
Brief Title: Randomized-controlled Trial of Preoperative Inspiratory Muscle Training on Postoperative Complications
Acronym: INSPIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Lunge Zuerich (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-PreopInsp
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Complications; Breathing Exercises; Preoperative Period
Keywords: inspiratory muscle training; CCI; postoperative complications; prehabilitation; preoperative respiratory training
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Prospective randomized-controlled single-center trial, non-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training arm (Experimental): Patients perform inspiratory muscle training containing of 30 breaths twice a day for 14-18 days before surgery.
  Interventions: Behavioral: preoperative inspiratory muscle training
- Control arm (No Intervention): No preoperative inspiratory muscle training

INTERVENTIONS:
Behavioral: preoperative inspiratory muscle training — Physiotherapists will measure the maximal inspiration pressure (MIP) with the POWER®breathe device of each single patient. Patients will then be instructed to perform inspiratory muscle training at the level of 60% of their individual MIP. Patients are instructed to perform the training containing of 30 breaths twice a day for 14-18 days before surgery. The devices are able to register the performance of each single training session and training results are monitored.
  Arms: Training arm

SUMMARY:
Rehabilitation strategies after abdominal surgery enhance recovery and improve outcome. A cornerstone of rehabilitation is respiratory physiotherapy with inspiratory muscle training to enhance pulmonary function. Prehabilitation is the process of enhancing functional capacity before surgery in order to compensate for the stress of surgery and postoperative recovery. There is growing interest in deploying pre-habilitation interventions prior to surgery.

The aim of this study is to assess the impact of preoperative inspiratory muscle training on postoperative overall morbidity. The question is, whether inspiratory muscle training prior to elective abdominal surgery reduces the number of postoperative complications and their severity grade.

DETAILED DESCRIPTION:
INSPIRA is a prospective randomized-controlled single-center trial, non-blinded The aim of this study is to assess the impact of preoperative inspiratory muscle training on postoperative overall morbidity. The question is, whether inspiratory muscle training prior to elective abdominal surgery reduces the number of post-operative complications and their severity grade.

Furthermore, the impact of preoperative inspiratory muscle training on postoperative physiotherapeutic performance as surrogate of convalescence is assessed, too.

Patients will be instructed by physiotherapists to perform inspiratory muscle training containing of 30 breaths twice a day for 14-18 days before surgery using Power®Breathe KHP2.

Primary outcome is Comprehensive Complication Index (CCI) at 90 days after surgery. The CCI expresses morbidity on a con-tinuous numeric scale from 0 (no complication) to 100 (death) by weighing all postoperative complications according to the Clavien-Dindo classification for their respective severity.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Patient Informed Consent Form)
* Planned abdominal surgery with planned duration >2hours (disease localization: upper vs. lower gastro intestinal, HPB, hernia, others)
* Planned surgery at least two weeks after inclusion at outpatient clinic
* Male and female patient over 18 years

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, of the participant
* Known or suspected non-compliance, drug or alcohol abuse,
* Previous enrolment into the current study
* Participation in another study with inspiratory muscle training within 30 days preceding or during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 90 days postoperative
  Postoperative complications measured by the comprehensive complication index (CCI) Com-prehensive Complication Index (CCI) 90 days after surgery. The CCI expresses postoperative morbidity on a continuous numeric scale from 0 (no complication) to 100 (death) by weighing all postoperative complications according to the validated Clavien-Dindo classification for their respective severity. It is measured at the end-of hospitalization and 90 days after surgery to include cases in which a readmission was necessary. Postoperative complications are gold standard in evaluation of quality of surgery as they directly reflect the procedures out-come and are most relevant for the patients.

SECONDARY OUTCOMES:
Postoperative morbidity | At the end of hospitalization and 90 days +/- 2 weeks postoperative
  Secondary endpoints are the postoperative morbidity along the classification of Clavien-Dindo at the end of hospitalization as well as 90 days +/- 2 weeks after surgery. This classification consists of five (1-5) severity grades. Grade 1 reflects minor complications, while grade 5 re-flects death. The classification is widely accepted and validated to report postoperative compli-cations.
Length of hospital stay (LOS) | 90 days postoperative
  Length of postoperative hospital stay
Readmission rate | 90 days postoperative
  Readmission rate as reflection of postoperative outcome.
Mortality | 90 days postoperative
  Mortality as reflection of postoperative outcome.
Maximum inspiratory pressure (MIP) | 5 days after surgery
  MIP is the most commonly used measure to evaluate inspiratory muscle strength. Very sensitive in detecting early respiratory muscle dysfunction, it allows for the assessment of ventilatory failure, restrictive lung disease and respirato-ry muscle strength and therefore represents a clinically meaningful trial endpoint.
Load | 5 days after surgery
  Load (cmH20) (LOAD) is a measure of resistance to inhalation, and represents the pressure generated in the airways due to the force of the inspiratory muscles during a training session. As the training load decays with increasing lung volume (in order to match the length tension characteristics of the inspiratory muscles), the load displayed corresponds to the resistance at the start of inhalation (i.e. at RV). A higher load result means that the patient is training their inspiratory muscles hard-er, leading to stronger muscles. Stronger inspiratory muscles will need to work less hard to cope with the demands of breathing, leading to reduced breathlessness
Power (Watt) | 5 days after surgery
  POWER is a measure of muscle performance which combines strength and speed of move-ment (Pressure x Flow). More powerful muscles will be more resistant to fatigue at a given level of work and therefore, breathlessness will be reduced. The value displayed is the average power for all breaths in a training session.
Sit-to-stand test | 5 days after surgery
  During the sit-to-stand test, the quantity [n] how often a patient can sit down on a chair and stand up during 60 seconds is noted. These values are evaluated at admission to hospital for surgery and 5 days after surgery.
Energy (Joule) | 5 days after surgery
  Breathing Energy) is a measure of the mechanical work (or effort) of breathing during your breathing training session. It is a result which combines the force exerted by your inspiratory muscles and the volume of air inhaled. The higher the value of breathing energy you attain, the longer and harder you have worked your inspiratory muscles.
Volume (l) | 5 days after surgery
  Lung volume refers to the volume of gas the lungs and it represents the functions of the respiratory muscles and the mechanics of the lung and chest .

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lisa Birrer, MD, Principal Investigator — UniversitätsSpital Zürich (USZ)
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birrer DL, Kuemmerli C, Obwegeser A, Liebi M, von Felten S, Pettersson K, Horisberger K. INSPIRA: study protocol for a randomized-controlled trial about the effect of spirometry-assisted preoperative inspiratory muscle training on postoperative complications in abdominal surgery. Trials. 2022 Jun 7;23(1):473. doi: 10.1186/s13063-022-06254-4. PMID 35672861
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/35672861/